CLINICAL TRIAL: NCT03879369
Title: Sexual Dysfunction in Female Patients With Adult Acne Vulgaris
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa A Ghallab, principal investigator, Assiut University
Other Study IDs: ST ACNE
Record Dates: First submitted 2019-03-11; First posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hormonal assay — LH , FSH and Free testosterone index (FTI) levels

SUMMARY:
Assessment of sexual dysfunction in adult females with acne vulgaris and its relation to other variables as quality of life, acne severity and hormonal dysfunction.

DETAILED DESCRIPTION:
Acne vulgaris is a common chronic inflammatory skin disease of pilosebaceous units. It is characterized by formation of comedones, erythematous papules, pustules and less frequently by nodules, deep pustules, or pseudocysts. In some cases, it may be accompanied by scarring. It is the most common dermatological condition affecting adolescents worldwide. It has a prevalence of almost 85% in people aged 12-24 years . Women have a high prevalence than men, especially after 25 years of age. It affects 12%-22% of women in their adult life.

Several factors are involved in the pathogenesis of the disease including abnormal sebum production, altered follicular keratinization with subsequent follicular plugging and Propionibacterium acnes colonization . Also, endocrine factor or androgens are considered a major factor involved in the pathogenesis of the disease. It probably results from an androgen excess or exacerbated response of the pilosebaceous unit to the normal circulating androgen levels.

Polycystic ovary syndrome (PCOS) is the most common endocrine disorder to affect women in their reproductive years. It is characterized by hyperandrogenism which results in a series of skin changes including hirsutism, acne, seborrhea and androgenetic alopecia.

Acne vulgaris causes profound negative psychological and social effects on the quality of life (QoL) of patients. It has a great impact on appearance which is linked with self-esteem and self-confidence. Factors that influence the psychological impact of acne include perceived sexual attractiveness, relationships with family and friends, judgments of others, stigmatization, stress, and fear of scarring.

Several researches concluded that body image is an important psychological factor in women sexual well-being. Female sexual dysfunction may associate certain dermatologic diseases as a result of its effect on self-esteem and psychological conditions.

Despite acne vulgaris is a common disease in adult females, little is published on its effect on female sexual function. The published studies were concerned with sexual dysfunction in males with acne vulgaris receiving isotretinoin, females with genital acne (acne inversa) or those with frank hormonal disturbances. None of these studies concluded whether female sexual dysfunction is impaired with acne vulgaris as a relation to its effect on psychological wellbeing or due to associated endocrine factors or other disease variables.

The Female Sexual Function Index (FSFI) is a widely used measurement tool to assess female sexual function. Arabic translation of the FSFI (ArFSFI) has been validated and can be used in the Egyptian population. It is reliable and easy to be understood by women and it is as good as the original FSFI in assessing female sexual function.

The dermatology life quality index (DLQI) is another questionnaire that assess the impact of dermatologic diseases on patient psychometry. It was the first dermatology-specific QOl instrument and to date is the most commonly used.

Acne severity of the patients will be evaluated by the global acne grading system (GAGS). The GAGS is an acne grading system developed by Doshi et al. It is a simple, accurate and fast method for the determination of severity of acne. It requires no special equipment and is relatively cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* adult female patients with acne vulgaris between 18-40 years old

Exclusion Criteria:

any disease affecting sexual function will be excluded like

* female genital mutilation.
* females with other major medical, endocrine and genital comorbidities or receiving medications that affect sexual function.
* females with frank psychological disturbances.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — adult female patients with acne vulgaris between 18-40 years old and control group of matched age and sex
Study Population: adult female patients with acne vulgaris between 18-40 years old and control group of matched age and sex
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of sexual function using FSFI questionnaire | 30 minutes
  Summation of the mean score of the six domains of the FSFI questionnaire

REFERENCES:
- [Background] El-Hamd MA, Nada EEA, Moustafa MA, Mahboob-Allah RA. Prevalence of acne vulgaris and its impact of the quality of life among secondary school-aged adolescents in Sohag Province, Upper Egypt. J Cosmet Dermatol. 2017 Sep;16(3):370-373. doi: 10.1111/jocd.12328. Epub 2017 Mar 2. PMID 28256050
- [Background] Rocha MA, Bagatin E. Adult-onset acne: prevalence, impact, and management challenges. Clin Cosmet Investig Dermatol. 2018 Feb 1;11:59-69. doi: 10.2147/CCID.S137794. eCollection 2018. PMID 29440921
- [Background] Ragab M, Hassan EM, Elneily D, Fathallah N. Association of interleukin-6 gene promoter polymorphism with acne vulgaris and its severity. Clin Exp Dermatol. 2019 Aug;44(6):637-642. doi: 10.1111/ced.13864. Epub 2019 Jan 16. PMID 30652337
- [Background] Romanska-Gocka K, Wozniak M, Kaczmarek-Skamira E, Zegarska B. Abnormal plasma lipids profile in women with post-adolescent acne. Postepy Dermatol Alergol. 2018 Dec;35(6):605-608. doi: 10.5114/ada.2018.77612. Epub 2018 Nov 13. PMID 30618529
- [Background] Nasiri Amiri F, Ramezani Tehrani F, Esmailzadeh S, Tohidi M, Azizi F, Basirat Z. Sexual function in women with polycystic ovary syndrome and their hormonal and clinical correlations. Int J Impot Res. 2018 Apr;30(2):54-61. doi: 10.1038/s41443-017-0006-2. Epub 2017 Dec 15. PMID 29242633
- [Background] Gowri BV, Chandravathi PL, Sindhu PS, Naidu KS. Correlation of Skin Changes with Hormonal Changes in Polycystic Ovarian Syndrome: A Cross-sectional Study Clinical Study. Indian J Dermatol. 2015 Jul-Aug;60(4):419. doi: 10.4103/0019-5154.160505. PMID 26288423
- [Background] Chernyshov PV, Zouboulis CC, Tomas-Aragones L, Jemec GB, Manolache L, Tzellos T, Sampogna F, Evers AWM, Dessinioti C, Marron SE, Bettoli V, van Cranenburgh OD, Svensson A, Liakou AI, Poot F, Szepietowski JC, Salek MS, Finlay AY. Quality of life measurement in acne. Position Paper of the European Academy of Dermatology and Venereology Task Forces on Quality of Life and Patient Oriented Outcomes and Acne, Rosacea and Hidradenitis Suppurativa. J Eur Acad Dermatol Venereol. 2018 Feb;32(2):194-208. doi: 10.1111/jdv.14585. Epub 2017 Oct 10. PMID 28898474
- [Background] Dreno B, Bagatin E, Blume-Peytavi U, Rocha M, Gollnick H. Female type of adult acne: Physiological and psychological considerations and management. J Dtsch Dermatol Ges. 2018 Oct;16(10):1185-1194. doi: 10.1111/ddg.13664. Epub 2018 Sep 24. PMID 30248242
- [Background] Sarhan D, Mohammed GF, Gomaa AH, Eyada MM. Female Genital Dialogues: Female Genital Self-Image, Sexual Dysfunction, and Quality of Life in Patients With Vitiligo With and Without Genital Affection. J Sex Marital Ther. 2016;42(3):267-76. doi: 10.1080/0092623X.2015.1010678. Epub 2015 Feb 4. PMID 25650731
- [Background] Hassanin AM, Ismail NN, El Guindi A, Sowailam HA. The emotional burden of chronic skin disease dominates physical factors among women, adversely affecting quality of life and sexual function. J Psychosom Res. 2018 Dec;115:53-57. doi: 10.1016/j.jpsychores.2018.10.011. Epub 2018 Oct 22. PMID 30470317
- [Background] Healy D, Le Noury J, Mangin D. Enduring sexual dysfunction after treatment with antidepressants, 5alpha-reductase inhibitors and isotretinoin: 300 cases. Int J Risk Saf Med. 2018;29(3-4):125-134. doi: 10.3233/JRS-180744. PMID 29733030
- [Background] Kurek A, Peters EM, Chanwangpong A, Sabat R, Sterry W, Schneider-Burrus S. Profound disturbances of sexual health in patients with acne inversa. J Am Acad Dermatol. 2012 Sep;67(3):422-8, 428.e1. doi: 10.1016/j.jaad.2011.10.024. Epub 2011 Dec 17. PMID 22182915
- [Background] Hevesi K, Meszaros V, Kovi Z, Marki G, Szabo M. Different Characteristics of the Female Sexual Function Index in a Sample of Sexually Active and Inactive Women. J Sex Med. 2017 Sep;14(9):1133-1141. doi: 10.1016/j.jsxm.2017.07.008. PMID 28859872
- [Background] Anis TH, Gheit SA, Saied HS, Al kherbash SA. Arabic translation of Female Sexual Function Index and validation in an Egyptian population. J Sex Med. 2011 Dec;8(12):3370-8. doi: 10.1111/j.1743-6109.2011.02471.x. Epub 2011 Oct 13. PMID 21995610
- [Background] Basra MK, Fenech R, Gatt RM, Salek MS, Finlay AY. The Dermatology Life Quality Index 1994-2007: a comprehensive review of validation data and clinical results. Br J Dermatol. 2008 Nov;159(5):997-1035. doi: 10.1111/j.1365-2133.2008.08832.x. Epub 2008 Sep 15. PMID 18795920
- [Background] Doshi A, Zaheer A, Stiller MJ. A comparison of current acne grading systems and proposal of a novel system. Int J Dermatol. 1997 Jun;36(6):416-8. doi: 10.1046/j.1365-4362.1997.00099.x. No abstract available. PMID 9248884